CLINICAL TRIAL: NCT07281105
Title: A Multi-Site, Randomized, Placebo-Controlled, Double-Blind, Phase 2 Clinical Trial of EG-501 for the Treatment of Cognitive Impairment in Systemic Lupus Erythematosus
Brief Title: EG-501 for Cognitive Impairment in Neuropsychiatric SLE (NPSLE): Efficacy and Safety Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evergreen Therapeutics, Inc. (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EG-501-2.1
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neuropsychiatric Systemic Lupus Erythematosus; Systemic Lupus Erythematosus (SLE); Cognitive Impairment
MeSH Terms: conditions — Lupus Vasculitis, Central Nervous System; Lupus Erythematosus, Systemic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Stratified, randomized, double-blind, placebo-controlled, parallel group study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Placebo (Placebo Comparator): At randomization, subjects will receive one matching placebo capsule twice per day for one week. One matching placebo capsule twice per day will be taken for the next week (Week 2), then one matching placebo capsule in the morning and two capsules at night for one week (Week 3), and finally two capsules twice per day for three weeks (Weeks 4-6). Maximum tolerated number of capsules will be determined at this time and this dose will be continued for an additional six weeks.
  Interventions: Drug: Placebo
- Drug: EG-501 (Experimental): EG-501/ EG-MNTP-01, Strength: 5 mg or 10 mg, oral capsules
  At randomization, subjects will receive 5 mg twice per day for one week. Dose will be escalated to 10 mg twice per day for one week, then 10 mg in the morning and 20 mg at night for one week, and finally 20 mg twice per day for three weeks. Maximum tolerated will be determined at this time and this dose will be continued for an additional six weeks.
  Interventions: Drug: EG-501

INTERVENTIONS:
Drug: Placebo — The placebo will match the study drug in appearance, dose, and frequency. It will not contain any active drug (EG-501).
  Arms: Drug: Placebo
Drug: EG-501 — EG-501/ EG-MNTP-01 is an oral, low-affinity NMDA receptor antagonist.
  Other Names: EG-MNTP-01
  Arms: Drug: EG-501

SUMMARY:
Neuropsychiatric systemic lupus erythematosus with cognitive impairment (NPSLE-CI) is a serious, disabling, and potentially life-threatening manifestation of SLE, affecting up to 80% of patients with cognitive impairments ("brain fog"), leading to substantial disability, approximately 2 times higher unemployment risk, reduced health-related quality of life (HRQoL), and mortality 2-14 times higher than the general population (standardized mortality ratio, SMR). No approved therapies exist for NPSLE cognitive dysfunction, representing a high-priority unmet need for this FDA-recognized serious condition with major functional and psychosocial burden. The objective of this study is to evaluate the safety, tolerability and efficacy of EG-501 in a precise patient subset with NPSLE. Participants will complete a full 14-week clinical trial, receiving either EG-501 or a placebo.

DETAILED DESCRIPTION:
Protocol EG-501-2.1 is a Phase 2, multi-site, randomized, double-blind, placebo-controlled trial evaluating the efficacy, safety, and tolerability of EG-501 for the treatment of cognitive impairment in systemic lupus erythematosus (SLE). The primary objective was to assess whether a 12-week EG-501 regimen produces a statistically and clinically significant improvement in the Total Scale Index score of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS®), compared with matched placebo, in a precisely defined SLE population with objective cognitive impairment. Fifty-six (56) patients were randomized treatment, 30 to placebo group and 26 to EG-501 group. All but three patients were female. Median age was 44.0 and 45.5 for placebo and EG-501 groups, respectively. With patients recruited only from the US, racial distribution was about 2/3 white, 1/3 black, with ethnicity reflecting largely non-Hispanic demographics.

ELIGIBILITY:
Key Inclusion Criteria:

1. Physician diagnosis of SLE;
2. Report NPSLE symptoms on the screening survey recommended by EULAR guideline but limited to a subset of the psychiatric manifestations questions and using a cut-off score of at least 5, with a minimum of 2.5 being scored on section 1;
3. Score ≤ 85 on the RBANS total index (≤ 1 SD below the normative mean of 100)

Key Exclusion Criteria:

1. Male and female subjects <18 or >69 years;
2. Change in medication that may affect mood or cognition including prednisone, antidepressant medications, analgesics including opioids, or stimulants within the last 4 weeks;
3. Metabolic derangement defined as liver function tests >3x upper limit of normal, or severe renal disease defined as calculated creatinine clearance<30 mL;
4. Severe psychiatric disease including schizophrenia, psychosis, suicidal depression, or substance abuse disorder;
5. Other factors which in the opinion of the investigator could potentially impact the study outcomes (e.g., underlying disease, medications, history)* or prevent the participant from completing the protocol (poor compliance or unpredictable schedule);

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Repeatable Battery for Assessment of Neuropsychological Status (RBANS) Total Index Score at endpoint (Visit 4) | 12 weeks
  RBANS is a widely used psychiatric tool that objectively measures cognitive impairment. It is comprised of 12 subtests and takes approximately 30 minutes. For scoring, the RBANS index scores are converted to classifications including Very Superior (130 and above), Superior (120-129), High Average (110-119), Average (90-109), Low Average (80-89), Borderline (70-79), and Extremely Low (69 and below). A score of Extremely Low equates to severe cognitive impairment.
  The primary outcome measure will be analyzed using ANCOVA controlling for EG-501 or placebo, baseline RBANS, sex, age, and NMDAR status.

SECONDARY OUTCOMES:
RBANS Subscales | 12 weeks
  Our primary outcome is the RBANS Total Index Score, which is the sum of several subscales/tests. For a secondary outcome, each subscale/test individually to see if there is a trend for any one test in particular will be recorded. The subscales are all scored the same (40 - 160) and include immediate memory, delayed memory, visuospatial/constructional, language, and attention.
Incidence of Treatment-Emergent Adverse Events | 12 weeks
  The safety of EG-501 as measured by treatment-emergent adverse events will be determined.
Polysymptomatic Distress Scale | 12 weeks
  The Polysymptomatic Distress (PSD) scale measures the effect of PSD over a range of pain-related clinical symptoms. The scale was derived from variables used in the 2010 American College of Rheumatology fibromyalgia criteria, modified for use in clinical research, and broadened to be applicable for patients not meeting fibromyalgia diagnostic criteria. The PSD score is calculated by summing two components, the Widespread Pain Index (WPI) and Symptom Severity Scale (SSS). The WPI is a count of painful nonarticular body regions, and the SSS is a symptom severity measure that includes fatigue, sleep, and cognitive problems.
Beck Depression Inventory | 12 weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-report inventory that measures depression symptoms and attitudes. It takes approximately 10 minutes to complete and requires a fifth to sixth grade reading level to adequately comprehend the questions.
Hospital Anxiety and Depression Scale | 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale and was developed to detect states of depression, anxiety, and emotional distress among patients who were being treated for a variety of clinical problems. The scale has a total of 14 items, with responses being scored on a scale of 0-3 (3 indicates higher symptom frequencies). Scores for each subscale (anxiety and depression) range from 0 to 21, categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21.
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K | 12 weeks
  SLEDAI-2K is an updated version of the SLEDAI which was originally developed in 1985 as a clinical index to assess lupus disease activity in the preceding 10 days. It is a cumulative and weighted index of 24 different clinical and laboratory variables/disease descriptors, comprising 9 organ systems. The Investigator will assess disease descriptors on the SLEDAI-2K collection sheet (e.g., arthritis, myositis, alopecia, rash, mucosal ulcers, etc.).
Patient Global Impression of Change (PGIC) | 12 weeks, Endpoint (Visit 4)
  Participants will answer the standard question, "Considering all the ways your health affects you, how are you doing since the beginning of your treatment?" Answers include very much worse, much worse, worse, unchanged, improved, much improved, and very much improved.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J. Crofford, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Health Houston, Houston, Texas